CLINICAL TRIAL: NCT03806751
Title: A Noninvasive Arterial Input Estimation Method for O-15 PET and Integrated PET/MR Scanning
Acronym: O-15 Water
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The investigator decided not to pursue the study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R18-010
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Validation of a New Noninvasive Method to Obtain the Arterial Input Function (AIF) Directly by PET Imaging
MeSH Terms: interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [O-15]water PET/MRI (Experimental): Volunteers will have two brain PET/MRI scans; first scan after injection of [O-15]water; second scan after injection of 1 gram of acetazolamide followed by injection of [O-15]water.
  Interventions: Drug: [O-15]Water; Drug: Acetazolamide

INTERVENTIONS:
Drug: [O-15]Water — All study participants with undergo brain imaging with [O-15]water-PET/MRI without and with administration of the carbonic anhydrase inhibitor acetazolamide. The PET tracer will be used to measure regional cerebral perfusion, and the administration of acetazolamide will lead to increased cerebral perfusion compared to baseline cerebral perfusion.
Drug: Acetazolamide — The administration of acetazolamide will lead to increased cerebral perfusion compared to baseline cerebral perfusion.
  Other Names: Diamox

SUMMARY:
The overall aim of this project is to implement a non-invasive method of measuring quantitative regional cerebral blood flow (rCBF) on the UAB hybrid PET/MRI scanner to allow conducting such [O-15]water based scans with relative ease and safety in a large variety of important clinical and research applications. Participants will undergo imaging at baseline and after administration of a drug to increase cerebral blood flow to evaluate perfusion estimates during low and high flow states. The goal of this study is to generate data that will justify eliminating invasive arterial sampling in most [O-15]water-based PET protocols.

ELIGIBILITY:
Inclusion Criteria:

* Six participants aged 19-60 years of age, male and female, with no evidence of neurological disease, will be recruited from UAB and the surrounding community.

Exclusion Criteria:

* Participants will be excluded if there is any evidence or history of claustrophobia or the subject has metallic implants or devices that are normally exclusion factors for MRI.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of arterial sampling to non-invasive methods to measure regional cerebral blood flow using [O-15]water-PET/MRI | 3 years
  Measurements of regional cerebral blood flow with [O-15]water-PET/MRI using arterial sampling versus non-invasive image-based input function estimates will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Advanced Imaging Facility, Birmingham, Alabama, United States